CLINICAL TRIAL: NCT01605331
Title: Safety and Efficacy of SR-hGH (Sustained-release Human Growth Hormone, Declage Inj.)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-SHCL007
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Growth Hormone Deficiency
Keywords: Adults; GH deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

ARMS (1):
- sustained-release recombinant human GH (SR-rhGH) (Experimental): 12-week subcutaneous administration, 2mg/week
  Interventions: Drug: sustained-release recombinant human GH (SR-rhGH)

INTERVENTIONS:
Drug: sustained-release recombinant human GH (SR-rhGH)

SUMMARY:
As studies demonstrate, the administration of recombinant human GH (rhGH) in adults with GH deficiency has been known to improve metabolic impairment and quality of life. Patients, however, do have to tolerate daily injections of GH (rhGH).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 20 years with diagnosed GH deficiency (caused by pituitary tumor, trauma, other pituitary disease)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety | 12 weeks
  Adverse event

SECONDARY OUTCOMES:
Efficacy | 12 weeks
  QoL-AGHDA